CLINICAL TRIAL: NCT06470048
Title: A Randomized, Double-blind, Parallel Group, Placebo-controlled Multicenter Study to Evaluate Efficacy, Safety and Tolerability of Ianalumab in Participants With Diffuse Cutaneous Systemic Sclerosis
Brief Title: A Clinical Study to Evaluate Ianalumab in Participants With Diffuse Cutaneous Systemic Sclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736S12201; 2024-511933-36-00 (Registry Identifier: EU CT number)
Expanded Access: NCT07244289 (Available)
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: Diffuse Cutaneous Systemic Sclerosis (dcSSc); Diffuse Scleroderma; Diffuse Systemic Sclerosis; Scleroderma, Diffuse; Scleroderma, Progressive; Sclerosis, Progressive Systemic; Sudden Onset Scleroderma; B cell depletion; Revised Composite Response Index in Systemic Sclerosis 25 (rCRISS25); modified Rodnan skin score; forced vital capacity
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAY736 (Ianalumab) (Experimental): Treatment Period 1:
  Ianalumab subcutaneous (s.c.) injection as defined in the protocol
  Treatment Period 2:
  Open-label (OL) Ianalumab subcutaneous (s.c.) injection as defined in the protocol
  Interventions: Drug: Ianalumab
- Placebo (Placebo Comparator): Treatment Period 1:
  Placebo to Ianalumab subcutaneous (s.c.) injection as defined in the protocol
  Treatment Period 2:
  Open-label (OL) Ianalumab subcutaneous (s.c.) injection as defined in the protocol
  Interventions: Drug: Placebo; Drug: Ianalumab

INTERVENTIONS:
Drug: Placebo — Ianalumab matching placebo subcutaneous (s.c.) injection as defined in the protocol
  Arms: Placebo
Drug: Ianalumab — subcutaneous (s.c.) injection as defined in the protocol
  Other Names: VAY736

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerability of s.c. ianalumab administered in participants with diffuse cutaneous systemic sclerosis relative to placebo

DETAILED DESCRIPTION:
The study consists of the following periods:

* Screening Period, with a duration of up to 6 weeks;
* Treatment Period 1, with a duration of 52 weeks;
* Treatment Period 2 (Open-label treatment), with a duration of 52 weeks;
* Post-treatment Follow-up Period, with a duration of at least 20 weeks post last dose and up to 2 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female participants >= 18 and =< 70 years (at the time of the screening visit).
* Diagnosis of systemic sclerosis, as defined by the 2013 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) classification criteria for SSc (van den Hoogen et al 2013) and meet the dcSSc subset classification according to LeRoy (LeRoy 1988)
* Disease duration of =< 60 months (defined as time from the first non-Raynaud phenomenon manifestation, e.g., puffy hands, scleroderma, digital ulcers, arthralgia, dyspnea)
* mRSS units of >= 15 and =< 45 at the time of the screening visit
* Active disease that meets at least one of the following criteria at screening:

  * Disease duration of =< 18 months defined as time from the first non-Raynaud phenomenon manifestation
  * Increase in mRSS of >= 3 units compared with the most recent assessment performed within the previous 6 months
  * Involvement of one new body area and an increase in mRSS of >= 2 units compared with the most recent assessment performed within the previous 6 months
  * Involvement of two new body areas within the previous 6 months
  * Elevated acute phase reactants (ESR) >= 30 mm/hr or high-sensitivity C-reactive protein (hsCRP) >= 6 mg/L)
  * Presence of SSc-interstitial lung disease (ILD) and ATA autoantibody positivity
  * Modified EUSTAR disease activity index (mDAI) ≥ 2.5
* Participant must be positive for at least one of the following autoantibodies:

  * anti-topoisomerase I (ATA) (also known as anti-SCL-70)
  * anti-RNA polymerase III (anti-RNAP3)
  * anti-nuclear antibody (ANA) (≥ 1:80) Participants who are positive only for ANA (while being negative for both ATA /anti-RNAP3) will be limited to 30% of the overall randomized study population.

Key Exclusion Criteria:

* Rheumatic disease other than dcSSc, including limited cutaneous disease (lcSSc) or sine scleroderma at the screening visit. Secondary Sjogren's disease and scleroderma myopathy are not exclusionary.
* Positive anti-centromere antibody (ACA+) without positive ATA or anti-RNAP3 autoantibody result at the screening visit
* Previous improvement (decrease) in mRSS > 10 units
* Pulmonary disease with FVC ≤ 50% of predicted or diffusing capacity of the lung for carbon monoxide (DLCO, corrected for hemoglobin) ≤ 40% of predicted at the screening visit
* WHO Functional Class 3 or higher assessment for pulmonary arterial hypertension (PAH, as defined on right heart catheterization), receiving IV therapy for PAH or evidence of other moderately severe pulmonary disease
* Participants treated with cyclophosphamide within 12 weeks prior to Baseline.
* Prior use of a B-cell depleting therapy other than ianalumab (e.g., rituximab, other anti-CD20 mAb, anti-CD22 mAb, or anti-CD52 mAb) administered within 36 weeks prior to randomization, or as long as B cell count is less than the lower limit of normal or baseline value prior to receipt of B cell-depleting therapy (whichever is lower).
* Treatment with biologic agents, such as intravenous immunoglobulin or monoclonal antibodies, including marketed drugs, within 12 weeks or 5 half-lives (whichever is longer) prior to baseline visit, unless explicitly allowed in inclusion criteria.
* Treatment with any investigational agent within ≤ 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of the baseline visit.
* Use of anti-fibrotic agents including colchicine, D-penicillamine, pirfenidone, or tyrosine kinase inhibitors (e.g., nintedanib, nilotinib, imatinib, dasatinib) in the 4 weeks prior to baseline visit. Patients with SSc-ILD requiring antifibrotics for management of ILD during the study, as per investigator judgement, should be excluded.
* Previous treatment with chlorambucil, bone marrow transplantation or total lymphoid irradiation.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant from menarche until becoming post-menopausal, unless they are using highly effective methods of contraception (failure rate < 1% per year) while taking study treatment and for 6 months after stopping study treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2030-07-15 (Estimated)

PRIMARY OUTCOMES:
3/5 rCRISS25 response | Week 52
  To demonstrate the superiority of ianalumab, compared to placebo, in achieving 3/5 Revised Composite Response Index in Systemic Sclerosis 25 (rCRISS25) response at Week 52

SECONDARY OUTCOMES:
Change from baseline in FVC% predicted at Week 52 | Week 52
  To demonstrate the superiority of ianalumab, compared to placebo, on change from baseline in percent-predicted forced vital capacity (FVC%) at Week 52
Change from baseline in mRSS at Week 52 | Week 52
  To demonstrate the superiority of ianalumab, compared to placebo, on change from baseline in modified Rodnan Skin Score (mRSS) at Week 52
Change from baseline in HAQ-DI at Week 52 | Week 52
  To demonstrate the superiority of ianalumab, compared to placebo, on change from baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 52
Ianalumab concentrations in serum during treatment and Follow-up Period | Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52, Week 64, Week 76, Week 88, Week 104, Week 108, Week 112, Week 116, Week 120, Week 124 and Week 208
  To assess the pharmacokinetics of ianalumab
Incidence and titer of anti-drug (ianalumab) antibodies (ADAs) in serum over time | Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 52, Week 64, Week 76, Week 88, Week 104, Week 124, Week 208
  To evaluate the immunogenicity of ianalumab
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 208
  The distribution of adverse events for ianalumab will be done via the analysis of frequencies for Adverse Event (AEs) and Serious Adverse Event (SAEs) through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (110):
- United States (15):
  - Arizona Arthritis and Rheumatology Research PLLC, Mesa, Arizona
  - UCLA, Los Angeles, California
  - Hoag Hospital, Newport Beach, California
  - Clinical Res Of W Florida, Clearwater, Florida
  - GNP Research, Cooper City, Florida
  - IRIS Research and Development, Plantation, Florida
  - Sarasota Arthritis Res Ctr, Sarasota, Florida
  - University of Chicago Hospitals, Chicago, Illinois
  - UMC New Orleans, New Orleans, Louisiana
  - Uni Of Michigan Health System, Ann Arbor, Michigan
  - Clinical Research Inst of MI, Saint Clair Shores, Michigan
  - West Tennessee Research Institute, Jackson, Tennessee
  - Arthritis and Rheumatology Ins, Allen, Texas
  - Novel Research LLC, Bellaire, Texas
  - Prolato Clinical Research Center, Houston, Texas
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, San Miguel de Tucumán
- Novartis Investigative Site, Graz, Austria
- Novartis Investigative Site, Leuven, Belgium
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Sao Jose Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- China (7):
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Tianjin
- Colombia (5):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
- France (8):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (3):
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
- Greece (2):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Athens
- Hungary (2):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
- India (5):
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, New Delhi
- Italy (8):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
- Japan (13):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Toyama
- Malaysia (2):
  - Novartis Investigative Site, Cheras, Kuala Lumpur
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Chihuahua City
- Poland (2):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Vila Nova de Gaia
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Salamanca
- Taiwan (4):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taoyuan District
- Thailand (2):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Ankara, Yenimahalle
- United Kingdom (3):
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, London
- Vietnam (2):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com